CLINICAL TRIAL: NCT01461304
Title: Dietary Therapy for Inherited Disorders of Energy Metabolism
Brief Title: Compassionate Use of Triheptanoin (C7) for Inherited Disorders of Energy Metabolism
Status: No longer available | Type: Expanded Access
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Professor of Pediatrics/Human Genetics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO08020019
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Very Long-chain acylCoA Dehydrogenase (VLCAD) Deficiency; Carnitine Palmitoyltransferase Deficiencies (CPT1, CPT2); Mitochondrial Trifunctional Protein Deficiency; Long-chain Hydroxyacyl-CoA Dehydrogenase Deficiency; Glycogen Storage Disorders; Pyruvate Carboxylase Deficiency Disease; ACYL-CoA DEHYDROGENASE FAMILY, MEMBER 9, DEFICIENCY of; Barth Syndrome
Keywords: fatty acid oxidation; triheptanoin; long-chain fatty acid oxidation disorders; LCHADD; VLCADD; CPT1; CPT2; TFP; Glycogen Storage Disorders; GSD; Pyruvate Carboxylase; PC; ACAD9; Barth
MeSH Terms: conditions — VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Pyruvate Carboxylase Deficiency Disease; Acyl-CoA Dehydrogenase Family, Member 9, Deficiency of; Barth Syndrome | interventions — triheptanoin

INTERVENTIONS:
Drug: triheptanoin — subjects will receive a modified diet containing triheptanoin (up to 2 grams/kg/24 hours; subjects who experience cardiomyopathy may receive doses up to 4 grams/kg/24 hours), or continued on their previously established triheptanoin dose; not to exceed RDA for fat, substituted for their MCT oil and/or natural fat. Study subjects will continue the triheptanoin-supplemented diet for a period of 12 months and then be able to continue into an indefinite extension phase in this compassionate use study. Laboratory evaluations will take place at two, six, and twelve months as well as every 12 months in the extension phase.
  Other Names: C7

SUMMARY:
This is a compassionate use study to allow patients already taking triheptanoin (C7) through previous studies to continue to receive the supplement. It will also allow triheptanoin supplementation in patients with qualifying disorders if they are failing conventional therapy.

DETAILED DESCRIPTION:
This study will treat children and adults who have documented deficiencies of mitochondrial fatty acid oxidation including disorders of the following enzymes: Carnitine-Acylcarnitine Translocase (CATR), Carnitine Palmitoyltransferase I and II (CPT I, CPT II), Very-Long Chain Acyl-CoA dehydrogenase (VLCAD), L-3-Hydroxy-Acyl-CoA Dehydrogenase (LCHAD), Acyl-CoA Dehydrogenase type 9 (ACAD9) and Mitochondrial Trifunctional Protein (TFP) with triheptanoin oil. This study is also open to patients with any type of glycogen storage disease, pyruvate carboxylase deficiency, or Barth Syndrome.

Symptoms often persist with standard diet including supplementation with medium chain triglyceride oil. Preliminary data shows triheptanoin to reverse many of the clinical symptoms not well controlled by standard diet.

On study entry, clinical and laboratory assessments will be carried out with the subject on their usual home diet. A complete history and physical exam will be performed. An echocardiogram must be obtained within the past year or it will be performed on the day of study entry. Following analysis of their diet and a negative pregnancy test, subjects will receive a modified diet containing triheptanoin (up to 2 grams/kg/24 hours for most subjects; subjects who experience cardiomyopathy may receive doses up to 4 grams/kg/24 hours), or continued on their previously established triheptanoin dose; not to exceed RDA for fat, substituted for their MCT oil and/or natural fat. This will be given by g-tube or orally divided into 2 or more doses. The dose will be adjusted on the basis of safety laboratory monitoring at specific time points and for adverse symptoms. The remainder of their diet will be modified to maintain appropriate caloric intake and balance. Total calories appropriate for RDA will be prescribed.

Study subjects will continue the triheptanoin-supplemented diet for a period of 12 months and then be able to continue into an indefinite extension phase in this compassionate use study. Laboratory evaluations will take place at two, six, and twelve months, as well as every 12 months in the extension phase. Laboratory tests may be completed at a local lab and the results forwarded to the PI for review between visits in Pittsburgh. Patients will monitor their weight at home on a monthly basis. Interim metabolic evaluations will be arranged as needed on a clinical basis with the study PI or the subject's home metabolic physician. Following the initial 12 months of the protocol, subjects will be placed on a continuing schedule for maintenance of triheptanoin therapy with a yearly follow up visit for an undeterminable period of time. Echocardiograms must be completed on an annual basis and sent to the study PI to review.

Travel to Pittsburgh, PA at the start of the study and annually is the responsibility of the subjects. Additionally, there may be study costs that insurance will not cover and subjects will be responsible for covering them. Examples of out-of-pocket study costs subjects may incur in addition to travel expenses including the following: necessary laboratory testing and echocardiograms. The study medication will be provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 month and up
* Diagnosis of disorder in long chain fatty acid oxidation, glycogen storage disease, pyruvate carboxylase deficiency, or Barth Syndrome
* Currently receiving triheptanoin as result of participation in previous study will be eligible if they have one of the included diagnoses
* Prefer 2 of following 3: acylcarnitine profile, fibroblast acylcarnitine profile or positive medical genetic test

Exclusion Criteria:

* Pregnant females
* MCAD deficiency
* disorder of short and medium chain fatty acid oxidation or ketone body metabolism

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Vockley, MD, PhD, Principal Investigator — Children's Hospital of Pittsburgh, University of Pittsburgh
Locations (1):
- University of Pittsburgh Division of Medical Genetics, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States